CLINICAL TRIAL: NCT05304728
Title: Sepsis Onset Warning System [SOWS] Master Enrollment Study Protocol
Brief Title: Sepsis Clinical Decision Support [CDS] Master Enrollment Study Protocol
Status: Enrolling by invitation | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2.7.2-1
Record Dates: First submitted 2022-03-23; First posted 2022-03-31 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Severe Sepsis; Severe Sepsis Without Septic Shock
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primary Objective: Severe Sepsis: The primary endpoint for this study is defined as the presence of sufficient data for SOWS training and algorithm development to proceed with subsequent validation. To provide sufficient data subsets (severe sepsis EHR encounters) for training and validation of the Sepsis Onset Warning System algorithm. There will not be any interventions administered.

SUMMARY:
This protocol will collect real-world data retrospectively from the electronic health record (EHR) as data obtained from the delivery of routine medical care to develop a machine learning (ML)-based Clinical Decision Support (CDS) system for severe sepsis prediction and detection.

DETAILED DESCRIPTION:
The purpose of this study is to gather data for the clinical development of the Sepsis Onset Warning System (SOWS) Software as Medical Device (SaMD) product to support a De Novo FDA submission and commercialization in the United States. Product development of SOWS is funded in part with federal funds from the Department of Health and Human Services; Office of the Assistant Secretary for Preparedness and Response; Biomedical Advanced Research and Development Authority.

Data will be obtained from passive prospective collection of patient encounter data throughout the duration of the planned study to support the product development life cycle activities associated with developing the Sepsis Onset Warning System (SOWS) for severe sepsis risk detection. Inputs from patient health records in combination with proprietary hematology parameters developed by Beckman Coulter, such as Monocyte Distribution Width (MDW), will be used. The SOWS tool will look to use clinical measurements which are commonly and reliably available in the EHR as structured data elements, such as heart rate, temperature, blood pressure, and laboratory results and account for changes in these values over time.

ELIGIBILITY:
Inclusion Criteria:

* All races, ages and ethnicities
* All patients admitted to the hospital or presenting to the Emergency Department

Exclusion Criteria:

* Patients not presenting to a hospital setting (e.g. urgent care, outpatient clinic excluded).

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This protocol has open enrollment to all genders, ages, and health statuses in patients admitted to the hospital or presenting to the ED.
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe Sepsis | Within 6 hours from presentation to the emergency department
  Identify patients having Severe Sepsis with the use of electronic health data

SECONDARY OUTCOMES:
Mortality | Within 6hours from presentation to the emergency department
  Hospital mortality at hospital for Severe Sepsis patients identified by algorithm using electronic health data as potential benefits for increased early detection of risk of severe sepsis
Length of Stay | Within 6hours from presentation to the emergency department
  Determine length of stay at hospital for Severe Sepsis patients identified by algorithm using electronic health data as potential benefits for increased early detection of risk of severe sepsis
Re-admission Rates | Within 6hours from presentation to the emergency department
  Determine potential reduction of hospital readmission rates for Severe Sepsis patients identified by algorithm using electronic health data as potential benefits for increased early detection of risk of severe sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Crouser, MD, Principal Investigator — Ohio State University
Locations (10):
- United States (10):
  - University of California, Irvine, Irvine, California
  - Augusta University Medical School, Augusta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - University Health/ Truman Medical Center, Kansas City, Missouri
  - University of Kansas Medical Center, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - WakeMed Health, Raleigh, North Carolina
  - University of Cininnati, Cincinnati, Ohio
  - MetroHealth Systems, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
Data elements will be retrospectively extracted from electronic health records from the respective sites and fed into the algorithm for performance testing. These data elements will not be shared with other researchers